CLINICAL TRIAL: NCT05268965
Title: Autonomic and Subjective Correlates of Affective Forecasting Skills in Post-traumatic Stress Disorder
Brief Title: Study of Affective Forecasting Skills in Post-traumatic Stress Disorder
Acronym: TRAUPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0385; 2021-A01582-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-02-07; First posted 2022-03-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Emotion; Post-traumatic stress disorder; Affective forecasting; Virtual reality; Autonomic nervous system; Electrodermal activity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients meeting DSM-5 criteria for PTSD.
  Interventions: Behavioral: Experimental: group comparison
- Group 2: Healthy controls who experienced a traumatic event but did not meet DSM-5 criteria for PTSD
  Interventions: Behavioral: Experimental: group comparison
- Group 3: Healthy controls who did not experience a traumatic event
  Interventions: Behavioral: Experimental: group comparison

INTERVENTIONS:
Behavioral: Experimental: group comparison — * Standardized psychiatric interview (Mini International Neuropsychiatric Interview MINI)
  * State-Trait-Anxiety Inventory (Spielberger, 1993)
  * Beck Depression Inventory (BDI-II, 1998)
  * Cognitive Emotional Regulation Questionnaire (Jermann & al., 2006) Participant installation and testing: 2 stages (forecasting on a computer, and exposure in virtual reality)
  Task / affective forecasting:
  * Step 1: forecasting about one's own emotional responses regarding pleasant, neutral and unpleasant scenarios
  * Step 2: experience of the same scenarios in virtual reality

SUMMARY:
Post-traumatic stress disorder (PTSD) is associated with a marked tendency to have exaggerated and persistent negative beliefs and expectations about oneself or the world . Although posttraumatic stress symptoms have been shown to be associated with a tendency to negatively anticipate the future, affective forecasting skills (i.e., the ability to predict one's own emotional reactions in response to a future event) have never been explored in PTSD . The hypothesis that the PTSD is associated with a negative affective forecasting bias, characterized by a tendency to predict more intense emotional responses to future negative events.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and being able to express themselves in French
* Understanding of informed consent and signature of the study participation form
* Giving informed, dated and signed consent
* Benefiting from health insurance coverage
* Normal or corrected visual and auditory acuity to achieve normality
* Group 1 : DSM-5 PTSD criteria, assessed using CAPS and PTSD Checklist for DSM-5 (PCL-5, Weathers & al., 2013)
* Group 2: PTSD Criteria A only

Exclusion Criteria:

Refusal of participation after clear and fair information on the study.

* Visual or auditory sensory disability to participate in the study.
* Personal history of neurological disease or current neurological disease.
* Personal history of current psychiatric disorder or psychiatric disorder (excluding PTSD in patients in the experimental group), assessed via the MINI.
* Pregnant or breastfeeding women
* Consumption of toxic substances other than tobacco and alcohol.
* Minors or adults under guardianship, under judicial protection, persons deprived of liberty.
* Groups 2 and 3: personal history of psychiatric disorder or current psychiatric disorder and taking psychotropic drugs
* Group 1: personal history of psychiatric disorders or current psychiatric disorders other than anxiety, depressive, trauma and stress-related disorders and treatment with psychotropic drugs not stabilized

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: subjects suffering from post-traumatic stress disorder (PTSD)
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
difference of arousal assessments measured using the Self-Assessment Manikin between the prediction and emotional experience phases | During the experimental task (2 hours)
  To compare the subjective affective forecasting bias between the PTSD group and the two control groups

SECONDARY OUTCOMES:
subjective correlates of the affective forecasting bias associated with PTSD changes in: valence scores. | During the experimental task (2 hours)
  valence scores using the Self-Assessment Manikin (Likert-type scale ranging from 1 [very unpleasant] to 9 [very pleasant])
autonomic correlates of the affective prediction bias associated with PTSD: changes in the skin conductance response and heart rate. | During the experimental task (2 hours)
  changes in the skin conductance response and heart rate assessed using a BIOPAC (System, inc).
link between PTSD symptomatology and affective forecasting bias | During the experimental task (2 hours)
  PTSD symptomatology assessed using the Clinician-Administered PTSD Scale (CAPS-5) and PTSD Checklist for DSM-5 (PCL-5)
link and correlation coefficients between biases measured at the neurovegetative (changes in heart rate and skin conductance) and subjective levels (arousal and valence ratings from the Self-Assessment Manikin) in PTSD | During the experimental task (2 hours)
link and correlation coefficients between affective forecasting bias and emotion regulation skills within each group | During the experimental task (2 hours)
  affective forecasting bias and emotion regulation skills, assessed using the Cognitive Emotional Regulation Questionnaire (CERQ)
link and correlation coefficients between affective forecasting bias and anxiety and depression | During the experimental task (2 hours)
  anxiety and depression, respectively assessed using the State-Trait-Anxiety Inventory (STAI) and the Beck Depression Inventory (BDI-II), within each group

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Vaiva, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Usn Fontan - Linquette Chu Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No